CLINICAL TRIAL: NCT05535296
Title: Prevention of Lifestyle-related Ill-health With Early Examinations of Health and Function and Individualized Risk Profiles (PREFUNKTION), a Pilot Study.
Brief Title: Prevention of Lifestyle-related Ill-health With Early Functional Examinations and Individualized Risk Profiles
Acronym: PREVFUNKTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lena Bornhoft (Other)
Collaborators: Vastra Gotaland Region (Other Government); Region Värmland, Sweden (Unknown)
Responsible Party: Sponsor-Investigator, Lena Bornhoft, Physiotherapist, PhD, Göteborg University
Organization: Göteborg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VGFOUREG-968488
Record Dates: First submitted 2022-08-30; First posted 2022-09-10 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Lifestyle Risk Reduction
Keywords: Prevention; Lifesyle-related condition; Physical function; Physical activity
MeSH Terms: conditions — Risk Reduction Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Standard health examination and related feedback. Functional examination. Risk profile and related advice.
  Interventions: Behavioral: Risk profile
- Control group (No Intervention): Standard health examination and related feedback. Functional examination.

INTERVENTIONS:
Behavioral: Risk profile — Compiliation of risk profile based on fitness, strength, mobility, balance, posture, physical activity level, weight and pain. Advice based on the above and support in goal-setting.
  Arms: Intervention group

SUMMARY:
Background: Many lifestyle-related health disorders are influenced by physical activity level and physical function. Health examinations which focus on musculoskeletal function of people who have risk factors for lifestyle-related disorders, combined with person-centered advice based on risk profiles can give people knowledge and guidance to manage their own lifestyle priorities.

Aim: To investigate the feasibility of a protocol for a randomized controlled trial (RCT) which will examine the preventive effects of musculoskeletal function examinations and person-centered advice on inactive middle-aged people.

Methods: Physically inactive middle-aged people will be invited to participate in a two-part health examination with follow-up after three months in a pilot study. Part 1 is a standard health examination including blood tests and Part 2 is a functional examination of fitness, strength, mobility, balance and posture according to our protocol based on validated tests. The intervention group receives feedback based on both parts of the examination while the control group receives feedback only from Part 1. Physical activity level will be measured objectively with accelerometers at inclusion and follow-up.

Expected results: The pilot study is expected to show whether the planned RCT is practically feasible and to give relevant support for the power analysis for a later full-scale RCT. Better understanding of personal physical function and risk factors can facilitate lifestyle decisions on the individual level which can reduce the risk for later ill-health and need of health-care. Preventive interventions may contribute to reduce the ever-increasing level of lifestyle-related ill-health.

ELIGIBILITY:
Inclusion Criteria:

* Born 1982 (aged 40 years). Self-assessed as physically inactive. Self-reported normal general mobility - can walk without support and has full use of all 4 extremities.

Exclusion Criteria:

* Self-reported regular moderate-to-intensive physical activity more than once per week. Pregnancy. Ongoing treatment requiring hospital-based services. Severe mental illness or intellectual impairment. Need of interpreter to participate in the study or answer the questionnaires.

Ages: 39 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Physical activity level | Change between inclusion and 3-4 month follow-up.
  Mean number of daily minutes in moderate-to-intensive physical activity measured with accelerometers during one week.
Participant feedback | Measured at 3-4 month follow-up.
  Rating of overall helpfulness of intervention in intervention group on 0 to 5 numerical rating scale ranging between 0=No help at all and 5=Very helpful.

SECONDARY OUTCOMES:
Participant feedback functional tests-Borg inclusion | Measured at inclusion.
  Rating of difficulty of individual functional tests on the Borg Rating of Perceived Exertion scale, ranging from 6 to 20 with higher levels indicating higher exertion level.
Participant feedback functional tests-Borg follow-up | Measured at 3-4 month follow-up.
  Rating of difficulty of individual functional tests on the Borg Rating of Perceived Exertion scale, ranging from 6 to 20 with higher levels indicating higher exertion level.
Participant feedback functional tests-instructions | Measured at inclusion.
  Rating of how understandable the instructions were on a 0 to 5 numerical rating scale where 0 is completely ununderstandable and 5 is very easy to understand.
Participant feedback - descriptive inclusion | Recorded at inclusion.
  Voluntary subjective impressions of the intervention
Participant feedback - descriptive follow-up | Recorded at 3-4 month follow-up.
  Voluntary subjective impressions of the intervention
Risk levels | Change between inclusion and 3-4 month follow-up.
  Change in risk levels on the risk profile.
Goal achievement | 3-4 month follow-up
  Proportion of goals set at inclusion achieved.
Ekblom-Bak fitness test | Change between inclusion and 3-4 month follow-up.
  Measured as VO2-max in ml/kg/min where higher values indicate better fitness level.
2-minute step test | Change between inclusion and 3-4 month follow-up.
  Measured with number of steps, where higher values indicate better fitness level.
Body mass index | Change between inclusion and 3-4 month follow-up.
  Calculated by weight in kg divided by squared height in meters.
Waist circumference | Change between inclusion and 3-4 month follow-up.
  Measured in centimeters with measuring tape.
Handgrip strength | Change between inclusion and 3-4 month follow-up.
  Measured with Jamar dynamometer, with higher numbers indicating greater strength.
30-second biceps test | Change between inclusion and 3-4 month follow-up.
  Measured by maximum number of repetitions with 2 kg (women) or 4 kg (men) dumbbell during 30 seconds, with higher numbers indicating greater strength.
Unilateral heel rise test | Change between inclusion and 3-4 month follow-up.
  Measured with maximum number of repetitions per leg, with higher numbers indicating greater strength.
30-second chair stand test | Change between inclusion and 3-4 month follow-up.
  Measured with maximum number of repetitions during 30 seconds, with higher numbers indicating greater strength.
Plank test | Change between inclusion and 3-4 month follow-up.
  Measured with maximum endurance time, with longer time indicating better trunk strength.
Sorenson's back extension test | Change between inclusion and 3-4 month follow-up.
  Measured with maximum endurance time, with longer time indicating better trunk strength.
Supine bridge test | Change between inclusion and 3-4 month follow-up.
  Measured with maximum endurance time, with longer time indicating better trunk strength.
Stand-on-one-leg eyes-open test | Change between inclusion and 3-4 month follow-up.
  Measured with maximum endurance time, with higher numbers indicating better balance.
Stand-on-one-leg eyes-closed test | Change between inclusion and 3-4 month follow-up.
  Measured with maximum endurance time, with higher numbers indicating better balance.
Sharpened Romberg | Change between inclusion and 3-4 month follow-up.
  Measured with maximum endurance time, with higher numbers indicating better balance.
Functional Reach test | Change between inclusion and 3-4 month follow-up.
  Measured with reach limit in centimeters, with higher numbers indicating better balance.
Lateral Reach test | Change between inclusion and 3-4 month follow-up.
  Measured with reach limit in centimeters, with higher numbers indicating better balance.
Navicular Drop test | Change between inclusion and 3-4 month follow-up.
  Measured as drop distance in millimeters, with higher numbers indicating higher dgree of pronation.
Occiput-to-wall test | Change between inclusion and 3-4 month follow-up.
  Measured as contact or no contact between head and wall.
Patella mobility | Change between inclusion and 3-4 month follow-up.
  Measured as locked or not locked patella in habitual standing position.
Sit-rise test | Change between inclusion and 3-4 month follow-up.
  Measured as points on 0-10 scale, with higher numbers indicating better mobility.
Fingertip-floor test | Change between inclusion and 3-4 month follow-up.
  Measured as distance in centimeters, with higher numbers indicating lower mobility.
Lateral flexion test | Change between inclusion and 3-4 month follow-up.
  Measured as distance in millimeters, with higher numbers indicating better mobility.
Beighton's hypermobility score | Measured at inclusion.
  Measured on 0 to 9 scale with higher numbers indicating higher level of hypermobility
Number of pain locations | Change between inclusion and 3-4 month follow-up.
  Change in number of pain locations on pain diagram.
Health-related quality of life | Change between inclusion and 3-4 month follow-up.
  Measured with Euroqol-5 dimensions, 5 questions and 0-100 barometer. Higher scores indicate better quality of life.
Self-reported physical activity_SGPALS | Change between inclusion and 3-4 month follow-up.
  Measured with Saltin-Grimby Physical Activity Level Scale (0 to 4 descriptive levels). Higher levels indicate more physically active.
Self-reported physical activity_SNBHW | Change between inclusion and 3-4 month follow-up.
  Measured with the Swedish National Board of Health and Welfare's 2 questions on physical activity (choose from 6 descriptive levels of exercise and 7 descriptive levels of daily activity). Higher levels indicate more physically active.
Sedentary time | Change between inclusion and 3-4 month follow-up.
  Measured with the SED-GIH question on time sitting still (7 levels from almost always to never). Higher levels indicate more physically active.
Risk for developing long-term musculoskeletal disorders | Change between inclusion and 3-4 month follow-up.
  Measured with the Örebro Musculoskeletal Pain Screening Questionnaire (10 questions, max 100 points, higher values indicate increased risk for longterm pain.
Blood pressure | Change between inclusion and 3-4 month follow-up.
  Change in blood pressure.
Blood tests | Change between inclusion and 3-4 month follow-up.
  Whether or not acceptable levels of serum cholesterol (3.3 to 6.9mmol/L), triglycerides (0.45 to 2.6 mmol/L), LDL-cholesterol (1.4 to 4.7 mmol/L), HDL cholesterol (women 1.0 to 2.7 and men 0.80 to 2.1 mmol/L) and blood glucose (4.0 to 6.0 mmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Lena Bornhöft, PhD, Principal Investigator — Region Västra Götaland, University of Gothenburg
Locations (1):
- Närhälsan Biskopsgården Health centre, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers than the participating research group.

REFERENCES:
- [Derived] Bornhoft L, Arvidsson D, Bergenheim A, Borjesson M, Fridolfsson J, Hellgren M, Nordeman L, Larsson MEH. Function-based risk reduction intervention for lifestyle-related disorders among inactive 40-year-old people: a pilot randomised controlled trial. BMC Public Health. 2024 Oct 13;24(1):2799. doi: 10.1186/s12889-024-20301-6. PMID 39396984
- [Derived] Bornhoft L, Arvidsson D, Bergenheim A, Borjesson M, Fridolfsson J, Hellgren M, Nordeman L, Larsson ME. Development and feasibility of a function-based preventive intervention for lifestyle-related disorders. BMC Public Health. 2024 Mar 4;24(1):681. doi: 10.1186/s12889-024-18017-8. PMID 38438859